CLINICAL TRIAL: NCT02264561
Title: The Effect of Caffeine on Attention
Brief Title: Caffeine's Effect on Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 14.12.NRC
Record Dates: First submitted 2014-09-24; First posted 2014-10-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Attention
MeSH Terms: interventions — Food; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Mannitol administered at visit 1 and at visit 2
  Interventions: Other: Food
- caffeine (Active Comparator): caffeine administered at visit 1 and at visit 2
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Active group
  Other Names: Caffeine
Other: Food — Control group
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine whether caffeine improves attention.

DETAILED DESCRIPTION:
Single centre single dose cross-over, placebo-controlled, double blind, randomized trial with two treatment conditions : caffeine and placebo

ELIGIBILITY:
Healthy male and female Aged 40-60 years

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Attention test: milliseconds and index of stimulus sensitivity | duration 10 days from screening to last visit (V2)

SECONDARY OUTCOMES:
Central Nervous System :response time. | duration: 10 days from screening to last visit (V2)
Mood measures: Visual Analog scale. | duration 10 days from screening to last visit V2

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Drug Research, Leiden, CL, Netherlands